CLINICAL TRIAL: NCT01591811
Title: Prospective Trial of Two Prone Breast Radiotherapy Techniques With Randomization to Concurrent Versus Weekly Boost
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-01299
Record Dates: First submitted 2012-04-26; First posted 2012-05-04 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Daily Boost of Radiation Therapy (Experimental): Arm 1 of treatment, you will be receiving 15 daily radiation fractions of 2.7 Gy (measure of radiation dose) daily for three weeks to the entire breast with a daily concomitant boost of 0.5 Gy
  Interventions: Radiation: Arm 1 Daily Boost of Radiation Therapy
- Arm 2 Weekly Boost of Radiation Therapy (Experimental): Arm 2 Weekly Boost will receive 15 daily radiation fractions of 2.7 Gy for three weeks to the entire breast with a weekly boost of 2.0 GY.
  Interventions: Radiation: Arm 2 Weekly Boost of Radiation Therapy

INTERVENTIONS:
Radiation: Arm 1 Daily Boost of Radiation Therapy — Arm 1 Daily boost. IMRT at 2.7Gy x15 fractions. Total dose 40.50Gy. Daily Boost 0.5Gy to tumor bed x 15 fractions. Tumor Bed Total=48Gy
  Other Names: Radiation Therapy
  Arms: Arm 1 Daily Boost of Radiation Therapy
Radiation: Arm 2 Weekly Boost of Radiation Therapy — Arm2: IMRT at 2.7Gy x 15 fractions. Total Dose=40.50 Gy. Weekly Boost 2Gy (on Friday). Tumor Bed Total 46.50Gy
  Other Names: Radiotherapy
  Arms: Arm 2 Weekly Boost of Radiation Therapy

SUMMARY:
1. To test the hypothesis that when prone, patients treated with 3D-CRT breast radiotherapy and randomly assigned to either a weekly or a daily boost to the tumor bed develop acute toxicity that is not significantly worse than that of a concurrent cohort of patients treated with IMRT randomly assigned to a weekly or daily boost regimen.
2. To test the hypothesis that when prone, patients treated with 3D-CRT breast radiotherapy, randomly assigned to either a weekly or a daily boost to the tumor bed develop late toxicity that is not significantly worse than that of concurrent cohort of patients treated with IMRT randomly assigned to a weekly of daily boost.
3. To test hypothesis that 5 year local control rates of ≤ 5% in-breast recurrence can be achieved in each of the two randomized arms, for either technique tested.

DETAILED DESCRIPTION:
During the past ten years the Breast Cancer Radiotherapy Research team at NYU has conducted a series of consecutive studies to optimize the safe delivery of accelerated radiotherapy to partial and whole breast in the prone position, as summarized in a recent review of this experience. The current protocol focuses on whole breast radiotherapy for women with stage 0-2 breast cancer treated by segmental mastectomy: it aims at further refining the role of prone IMRT versus a 3D-conformal radiotherapy technique in this common subset of patients.

This study is an open label randomized trial. Patients will be randomized within cohort defined by assigned treatment (3D CRT if IMRT not covered or IMRT) and within these primary strata by menopausal status (pre/post) and by chemotherapy prior to radiation (yes/no). The on-site treatment randomization assignments will done on site and treatment assignments will be provided to the Research Nurse after she has confirmed eligibility. Patients will be randomized within the primary strata based on presumed insurance coverage on consent to the study to allow simulation to proceed. Should the coverage change, then the patient will be re-randomized in the correct stratum and the initial randomization number will be retired with a notation that the initial stratification was revised and patient re-randomized.

Patients will have completed all breast surgical procedures prior to accrual into this protocol in order to establish eligibility criteria. Final pathology margins must be at least 1 mm in all directions to be eligible. The patient may undergo re-excision if the initial margins are involved or close (< 1mm). If the patient meets the eligibility criteria after re-excision, she may be entered onto the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or post-menopausal women with Stage 0, I and II breast cancer (Post-menopausal women defined as either (a) at least 2 years without menstrual period or (b) or patients older than 50 with serological evidence of post-menopausal status or (c) hysterectomized patients of any age with FSH confirmation of post-menopausal status)
2. Biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm
3. Status post segmental mastectomy, after sentinel node biopsy and/or axillary node dissection (DCIS and Tumors <5 mm in size do not require nodal assessment)
4. At least 2 weeks from last chemotherapy
5. Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

Exclusion Criteria:

1. Previous radiation therapy to the ipsilateral breast
2. More than 3 involved nodes identified at axillary staging, requiring adjuvant axillary radiation
3. Active connective tissue disorders, such as lupus or scleroderma
4. Prior or concurrent malignancy other than basal or squamous cell skin cancer or carcinoma in-situ of the cervix, unless disease-free > 3 years
5. Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute radiation toxicity of Grade 2 or higher. | Up to 90 days of radiation treatment
  By accruing 1000 patients randomized in strata defined by the two approaches to either weekly or daily boost, we will be able to establish the feasibility using different techniques and toxicity of prone breast radiotherapy with a weekly versus a daily boost, with IMRT and with 3DCRT non-IMRT approaches.
Number of patients with late radiation toxicity. | 90 days following radiation treatment up to 5years
  By accruing 1000 patients randomized in strata defined by the two approaches to either weekly or daily boost, we will be able to establish the feasibility using different techniques and toxicity of prone breast radiotherapy with a weekly versus a daily boost, with IMRT and with 3DCRT non-IMRT approaches.
Local Recurrence | up to 5 years
  To compare local control rates, distant recurrence and overall survival for weekly versus daily boost within strata defined by 3DCRT or IMRT at 2 and 5 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, M.D., Ph.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Cancer Institute, New York, New York, United States